CLINICAL TRIAL: NCT00960661
Title: A Randomized Trial Comparing Two Therapies: Basal Insulin/Glargine, Exenatide and Metformin Therapy (BET) or Basal Insulin/Glargine, Bolus Insulin Lispro and Metformin Therapy (BBT) in Subjects With Type 2 Diabetes Who Were Previously Treated by Basal Insulin Glargine With Either Metformin or Metformin and Sulfonylurea
Brief Title: A Trial Comparing Two Therapies: Basal Insulin/Glargine, Exenatide and Metformin Therapy (BET) or Basal Insulin/Glargine, Bolus Insulin Lispro and Metformin Therapy (BBT) in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-EW-GWDM
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; Byetta; insulin lispro; Humalog; insulin glargine; Lantus; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Insulin Lispro; Metformin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (BET) (Experimental): Basal Insulin/Glargine, Exenatide and Metformin Therapy (BET)
  Interventions: Drug: exenatide; Drug: Metformin; Drug: Insulin/ Glargine
- Insulin Lispro (BBT) (Active Comparator): Basal Insulin/Glargine, Bolus Insulin Lispro and Metformin Therapy (BBT)
  Interventions: Drug: insulin lispro; Drug: Metformin; Drug: Insulin/ Glargine

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg (4 weeks) followed by 10mcg (26 weeks), twice a day
  Other Names: Byetta
  Arms: Exenatide (BET)
Drug: insulin lispro — titrated based on pre-meal glucose level; three times a day
  Other Names: Humalog
  Arms: Insulin Lispro (BBT)
Drug: Metformin
Drug: Insulin/ Glargine

SUMMARY:
The study will compare two combination therapies: 1) Combined Basal Insulin Glargine (once a day), Exenatide (twice a day), and Metformin Therapy; or 2) Combined Basal Insulin Glargine (once a day), Bolus Insulin Lispro (three times a day), and Metformin Therapy, in subjects with Type 2 Diabetes Mellitus who have inadequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Have been taking a basal insulin Glargine, at dose of ≥ 20 units/day, for at least 3 months prior to study start.
* Have been taking basal insulin Glargine at dose of ≥ 20 units/day, in combination with 1 of the following oral antidiabetic medication (OAM) regimens, for at least 3 months prior to study start:

  * Metformin or immediate-release metformin or extended-release metformin alone at a maximum tolerated and stable dose with no less than 500 mg/day for at least 6 weeks prior to study start; or
  * Metformin or immediate-release metformin or extended-release metformin at a maximum tolerated and stable dose with no less than 500 mg/day for at least 6 weeks prior to study start and sulfonylurea at a stable dose for 6 weeks prior to study start.
* Have an HbA1C > 7.0% and ≤ 10.0%.
* Have a body mass index (BMI) between ≥ 25 and ≤ 45 kg/m2.

Exclusion Criteria:

* Are currently taking OAM that is not described above and not allowed with concurrent use of insulin per local product label.
* Have taken more than 1 week within 1 month prior to the study start any glucose-lowering medications not included above either alone or in combination formulations, or have used a drug for weight loss (for example, prescription drugs such as orlistat, sibutramine, phenylpropanolamine, rimonabant or similar over-the-counter medications).
* Have taken any insulin other than Glargine within the 3 months prior to study start for more than 1 week.
* Are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical, intraocular, and inhaled preparations) within 4 weeks prior to the study start.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device (other than the study drug/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have previously completed or been withdrawn from this study after enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (95):
- Argentina (8):
  - Research Site, Buenos Aires
  - Research Site, Caba
  - Research Site, Capital Federal
  - Research Site, Ciudad Autonoma de Buenos Aire
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Corrientes
  - Research Site, Rosario
  - Research Site, San Rafael
- Belgium (4):
  - Research Site, Arlon
  - Research Site, Bonheiden
  - Research Site, Edegem
  - Research Site, Merksem
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Oulu
  - Research Site, Vantaa
- France (16):
  - Research Site, Angers
  - Research Site, Auxerre
  - Research Site, Bar-le-Duc
  - Research Site, Douai
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochelle
  - Research Site, Le Creuzot
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nanterre
  - Research Site, Pessac
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Vénissieux
- Germany (8):
  - Research Site, Bad Lauterberg im Harz
  - Research Site, Dippoldiswalde
  - Research Site, Friedrichsthal
  - Research Site, Goch
  - Research Site, Grevenbroich
  - Research Site, Hamburg
  - Research Site, Mainz
  - Research Site, Saarbrücken
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Italy (6):
  - Research Site, Florence
  - Research Site, Napoli
  - Research Site, Olbia
  - Research Site, Perugia
  - Research Site, Trieste
  - Research Site, Verona
- Mexico (4):
  - Research Site, Aguascalientes
  - Research Site, Cuernavaca
  - Research Site, Mexico City
  - Research Site, Monterrey
- Netherlands (8):
  - Research Site, Almere Stad
  - Research Site, Amsterdam
  - Research Site, Beek
  - Research Site, Groningen
  - Research Site, Heerlen
  - Research Site, Hoogeveen
  - Research Site, Sittard-Geleen
  - Research Site, The Hague
- Portugal (3):
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Portugal
- Research Site, Hato Rey, Puerto Rico
- Romania (6):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Craiova
  - Research Site, Oradea
  - Research Site, Ploieşti
- Russia (3):
  - Research Site, Arkhangelsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
- South Korea (3):
  - Research Site, Seoul
  - Research Site, Ulsan
  - Research Site, Wŏnju
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Dos Hermanas
  - Research Site, Santander
  - Research Site, Valencia
- Sweden (7):
  - Research Site, Halmstad
  - Research Site, Karlstad
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Solna
  - Research Site, Stockholm
  - Research Site, Umeå
- United Kingdom (5):
  - Research Site, Bournemouth
  - Research Site, Ipswich
  - Research Site, Leicester
  - Research Site, Penarth
  - Research Site, Wakefield

REFERENCES:
- [Result] Diamant M, Nauck MA, Shaginian R, Malone JK, Cleall S, Reaney M, de Vries D, Hoogwerf BJ, MacConell L, Wolffenbuttel BH; 4B Study Group. Glucagon-like peptide 1 receptor agonist or bolus insulin with optimized basal insulin in type 2 diabetes. Diabetes Care. 2014 Oct;37(10):2763-73. doi: 10.2337/dc14-0876. Epub 2014 Jul 10. PMID 25011946

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1036 patients entered the study, 637 were assigned to the two interventional study groups. 10 patients assigned to treatment groups did not receive study drug.
Groups:
- Enrolled: Patients who enrolled in the basal insulin optimization (BIO) phase
Period: Basal Insulin Optimization Phase (BIO)
Arm/Group | Enrolled | Exenatide (BET) | Insulin Lispro (BBT)
Started | 1036 | 0 | 0
Completed | 637 | 0 | 0
Not Completed | 399 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Entry criteria not met | 331 | 0 | 0
Not completed — Withdrawal by Subject | 47 | 0 | 0
Not completed — Physician Decision | 8 | 0 | 0
Not completed — Sponsor decision | 3 | 0 | 0
Period: Interventional Phase
Arm/Group | Enrolled | Exenatide (BET) | Insulin Lispro (BBT)
Started | 0 | 316 | 321
Intent to Treat Population | 0 | 315 (all randomized participants who took at least one dose of study drug) | 312 (all randomized participants who took at least one dose of study drug)
Per Protocol Population | 0 | 247 (all randomized participants who completed study and had no violations) | 263 (all randomized participants who completed study and had no violations)
Completed | 0 | 264 | 275
Not Completed | 0 | 52 | 46
Not completed — Adverse Event | 0 | 17 | 8
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — entry criteria not met | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 7 | 2
Not completed — Withdrawal by Subject | 0 | 18 | 29
Not completed — Physician Decision | 0 | 3 | 5
Not completed — sponsor decision | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: per protocol population
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT) | Total
Number analyzed (Participants) | 247 | 263 | 510
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 180 | 182 | 362
  >=65 years | 67 | 81 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.6) | 59.4 (9.27) | 59.5 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 130 | 249
  Male | 128 | 133 | 261
prior use of Sulfonylurea (SU) [Number; unit: participants]
  YES | 85 | 99 | 184
  NO | 162 | 164 | 326
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent] | 8.27 (0.983) | 8.21 (0.871) | 8.24 (0.927)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c) From Baseline to Week 30
Description: Change in HbA1c from baseline following 30 weeks of therapy (i.e. HbA1c at week 30 minus HbA1c at baseline).
Time Frame: Baseline, 30 weeks
Population: Participants analyzed for this endpoint included the per protocol population, 247 and 263, respectively.
Measure: Least Squares Mean (Standard Error); unit: percent of hemoglobin
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 247 | 263
percent of hemoglobin | -1.13 (0.053) | -1.10 (0.051)
Statistical Analysis 1: Comparison: Exenatide (BET) vs Insulin Lispro (BBT); The primary objective is to test the hypothesis that BET is non inferior to BBT with respect to change in HbA1c from baseline to Week 30; Test type: Non-Inferiority or Equivalence — Non inferiority was concluded if the upper limit of the 95% confidence interval (CI) for the treatment contrast (BET minus BBT) at week 30 was less than the non inferiority margin; p = 0.6273, Mixed model repeated measures — The primary mixed-model repeated measures (MMRM) model included baseline HbA1c as covariate, treatment, country, prior use of SUs, week of visit, and treatment-by-week interaction as fixed effects and patient and error as random effects; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.18 to 0.11]

2. Secondary Outcome: Percentage of Participants Achieving HbA1C < 7.0%
Description: Percentage of participants achieving HbA1C < 7.0%
Time Frame: Week 30
Population: Participants included in the analysis = 244 and 263, respectively. These numbers derived from the per protocol population (247 and 263, respectively) with no missing data for this endpoint (244, 263, respectively).
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 244 | 263
Percentage of participants | 46.7 | 42.6

3. Secondary Outcome: Percent of Participants Achieving HbA1c ≤ 6.5%.
Description: Percent of participants achieving HbA1c ≤ 6.5%.
Time Frame: Week 30
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 244 | 263
percentage of participants | 26.2 | 25.5

4. Secondary Outcome: Change in Fasting Blood Glucose (FBG) From Baseline to Week 30.
Description: Change in fasting blood glucose (FBG) from Baseline to Week 30 using MMRM model. The model included the respective baseline outcome as covariate, treatment, country, prior use of SUs, week of visit, and treatment-by-week interaction as fixed effects and patient and error as random effects.
Time Frame: Baseline, Week 30
Population: Participants included in the analysis = 243 and 262, respectively. These numbers derived from the per protocol population (247 and 263, respectively) with no missing data for this endpoint (243, 262, respectively).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 243 | 262
mmol/L | -0.46 (0.155) | 0.18 (0.150)

5. Secondary Outcome: Change in Total Cholesterol From Baseline to Week 30
Description: Change in total cholesterol from baseline to Week 30 using ANCOVA model. The model included the respective secondary outcome as dependent variable, country, prior use of SU's and treatment groups as factors, and the respective outcomes baseline value as a covariate.
Time Frame: Baseline, week 30
Population: Participants included in the analysis = 237 and 254, respectively. These numbers derived from the per protocol population (247 and 263, respectively) with no missing data for this endpoint (237, 254, respectively).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 237 | 254
mmol/L | -0.14 (0.050) | -0.03 (0.049)

6. Secondary Outcome: Change in High Density Lipoprotein (HDL) From Baseline to Week 30
Description: Change in High Density Lipoprotein (HDL) from baseline to Week 30 using ANCOVA model.The model included the respective secondary outcome as dependent variable, country, prior use of SU's and treatment groups as factors, and the respective outcomes baseline value as a covariate.
Time Frame: Baseline, week 30
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 237 | 254
mmol/L | -0.04 (0.012) | 0.03 (0.012)

7. Secondary Outcome: Change in Low Density Lipoprotein (LDL) From Baseline to Week 30
Description: Change in Low Density Lipoprotein (LDL) from baseline to week 30 using ANCOVA model.The model included the respective secondary outcome as dependent variable, country, prior use of SU's and treatment groups as factors, and the respective outcomes baseline value as a covariate.
Time Frame: Baseline, Week 30
Population: Participants included in the analysis = 232 and 245, respectively. These numbers derived from the per protocol population (247 and 263, respectively) with no missing data for this endpoint (232, 245, respectively).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 232 | 245
mmol/L | -0.12 (0.042) | -0.03 (0.042)

8. Secondary Outcome: Change in Body Weight From Baseline to Week 30.
Description: Change in body weight from baseline to Week 30 using MMRM model.The model included the respective baseline outcome as covariate, treatment, country, prior use of SUs, week of visit, and treatment-by-week interaction as fixed effects and patient and error as random effects.
Time Frame: baseline, week 30
Population: Participants analyzed were 247 and 263, respectively. These were from the per protocol population (247, 263, respectively) with no missing data (247, 263, respectively).
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 247 | 263
kg | -2.45 (0.255) | 2.11 (0.247)

9. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 30
Description: Change in Systolic Blood Pressure (SBP) from baseline to Week 30 using MMRM model.The model included the respective baseline outcome as covariate, treatment, country, prior use of SUs, week of visit, and treatment-by-week interaction as fixed effects and patient and error as random effects.
Time Frame: Baseline, Week 30
Population: Participants included in the analysis = 207 and 227, respectively. These numbers derived from the per protocol population (247 and 263, respectively) with no missing data for this endpoint (207, 227, respectively).
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 207 | 227
mmHg | -4.13 (0.952) | 0.37 (0.919)

10. Secondary Outcome: Change in Diastolic Blood Pressure (DBP) From Baseline to Week 30
Description: Change in Diastolic Blood Pressure (DBP) from baseline to Week 30 using MMRM model.The model included the respective baseline outcome as covariate, treatment, country, prior use of SUs, week of visit, and treatment-by-week interaction as fixed effects and patient and error as random effects.
Time Frame: baseline, Week 30
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 207 | 227
mmHg | -0.64 (0.594) | -0.14 (0.572)

11. Secondary Outcome: Daily Insulin Glargine Dose at Baseline and at Week 30
Description: Daily Insulin Glargine Dose at baseline and at Week 30
Time Frame: Baseline, week 30
Population: Participants analyzed were from the per protocol population (247, 263) with no missing data for this endpoint (247, 263, respectively).
Measure: Mean (Standard Deviation); unit: IU/day
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 247 | 263
IU/day
  Baseline | 61.5 (30.94) | 61.1 (35.24)
  Week 30 | 56.9 (29.35) | 51.5 (31.44)

12. Secondary Outcome: Major Hypoglycemia Rate Per Year
Description: Mean (standard deviation) of major hyperglycemia episodes experienced per year. Rates per year were calculated for each individual as the number of episodes divided by the total number of days in the study (from randomization to last visit date), then multiplied by 365.25. Major hypoglycemia was defined as any symptoms consistent with hypoglycemia resulting in loss of consciousness or seizure that shows prompt recovery in response to administration of glucagon or glucose OR documented hypoglycemia (blood glucose <3.0 mmol/L [54 mg/dL]) and requiring the assistance of another person because of severe impairment in consciousness or behavior.
Time Frame: 30 weeks
Population: The As-treated population includes all randomized participants who had taken at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: rate per year
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 315 | 312
rate per year | 0.0 (0.23) [0 to 0] | 0.1 (0.39) [0 to 0]

13. Secondary Outcome: Minor Hypoglycemia Rate Per Year
Description: Mean (standard deviation) of minor hyperglycemia episodes experienced per year. Rates per year were calculated for each individual as the number of episodes divided by the total number of days in the study (from randomization to last visit date), then multiplied by 365.25. Minor hypoglycemia was defined as any time a participant feels that he or she is experiencing a sign or symptom associated with hypoglycemia that is either self-treated by the participant or resolves on its own AND has a concurrent finger stick blood glucose <3.0 mmol/L (54 mg/dL)
Time Frame: 30 weeks
Population: The As-treated population includes all randomized participants who had taken at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: rate per year
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Number analyzed (Participants) | 315 | 312
rate per year | 2.1 (5.08) [1.45 to 2.07] | 5.0 (12.83) [3.26 to 4.54]

ADVERSE EVENTS:
Description: As treated population, non-serious includes treatment emergent adverse events in both BIO (lead in) and intervention phases.
Arm/Group | Exenatide (BET) | Insulin Lispro (BBT)
Serious Adverse Events (participants affected / at risk) | 23/315 | 26/312
Other Adverse Events (participants affected / at risk) | 228/315 | 175/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (BET) (N=315) | Insulin Lispro (BBT) (N=312)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 2 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Post procedural infection (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Ureteroscopy (Investigations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery thrombosis (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial bypass operation (Surgical and medical procedures) | 0 | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (BET) (N=315) | Insulin Lispro (BBT) (N=312)
Diarrhoea (Gastrointestinal disorders) | 34 | 16
Dyspepsia (Gastrointestinal disorders) | 19 | 3
Nausea (Gastrointestinal disorders) | 102 | 5
Vomiting (Gastrointestinal disorders) | 39 | 3
Bronchitis (Infections and infestations) | 18 | 6
Influenza (Infections and infestations) | 18 | 16
Nasopharyngitis (Infections and infestations) | 37 | 20
Headache (Nervous system disorders) | 18 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 12 | 5
Decreased appetite (Metabolism and nutrition disorders) | 12 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 1
Urinary tract infection (Infections and infestations) | 11 | 7
Dizziness (Nervous system disorders) | 10 | 4
Pharyngitis (Infections and infestations) | 9 | 7
Gastroenteritis (Infections and infestations) | 8 | 2
Constipation (Gastrointestinal disorders) | 7 | 2
Gastritis (Gastrointestinal disorders) | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2
pain in extremity (General disorders) | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
seasonal allergy (Immune system disorders) | 5 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 9
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 7
upper respiratory tract infection (Infections and infestations) | 3 | 6
tooth infection (Infections and infestations) | 2 | 7
hypertension (Vascular disorders) | 2 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 5
anxiety (Psychiatric disorders) | 2 | 5
toothache (Gastrointestinal disorders) | 1 | 6
anemia (Blood and lymphatic system disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No